CLINICAL TRIAL: NCT01671072
Title: A Placebo Controlled, Single-blind, Randomized, Multi-center Phase 2B Study to Determine the Efficacy and Safety of TissueGene-C, an Allogeneic Human Chondrocytes Expressing TGF-b1, in Patients With Degenerative Arthritis
Brief Title: Efficacy and Safety Study of TissueGene-C to Degenerative Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kolon Life Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KS-TGC-01-2B
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Degenerative Arthritis
Keywords: Chondrocyte cells; Osteoarthritis; Gene therapy
MeSH Terms: conditions — Osteoarthritis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TissueGene-C (Experimental): Single intra-articular injection to the damaged knee joint a dose of 1.8 x 10^7 cells
  Interventions: Biological: TissueGene-C
- Normal Saline (Placebo Comparator): Single intra-articular injection to the damaged knee joint at the same volume
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: TissueGene-C — TissueGene-C at 1.8 x 10^7 cells
  Arms: TissueGene-C
Drug: Normal Saline — Sodium chloride 0.9%, 3.5ml
  Arms: Normal Saline

SUMMARY:
The purpose of this study is to determine whether TissueGene-C, an allogeneic human chondrocytes expressing Transforming Growth Factor(TGF)-b1, is effective and safe in patients with degenerative arthritis

DETAILED DESCRIPTION:
TissueGene-C is a biological new drug which consists of normal chondrocytes and transduced chondrocytes that express growth factors to regenerate the damaged cartilage tissues.

In the clinical trial Phase 2b, the investigators compared TissueGene-C to placebo during 6 - months trial with 54 outpatients who have had degenerative arthritis. The outpatients are assigned to TissueGene-C or placebo in 1:1 ratio, and will be monitored and recorded for improving clinical symptoms, sports activities, and function of the knee, and for the presence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Female or male aged 18 years or more
2. Diagnosed with degenerative arthritis of the knee
3. With an IKDC score of 60 or lower at the screening visit
4. With Grade 2 or 3 osteoarthritis as determined by the radiographic criteria of Kellgren and Lawrence
5. With a Body Mass Index(BMI) of higher than18.5 and lower than 30
6. With an International Cartilage Repair Society(ICRS) Grade IV cartilage damage in the major lesions, as confirmed through an MRI scan
7. With major lesions concentrated in one section of the knee, and with the major lesions considered the main cause of the clinical symptoms
8. With no alleviation of the symptoms even after at least three months of non-surgical treatment
9. Healthy, with no major findings from the physical examination, hematology, serum chemistry, and urine tests, and no significant medical history
10. Agreed to use an effective contraceptive method during the study period
11. Voluntarily agreed to participate in this study, and signed the informed consent form

Exclusion Criteria:

1. Showed clinically significant hematology, serum chemistry, and urine test results at the screening visit
2. Falls under Inclusion Criteria 6 but with the damage in the relevant lesion considered ICRS Grade IV sized more than 6 cm2
3. Took glucosamine, chondroitin, or any natural medicine within 14 days before the injection of the investigational product (but if the 14-day washout period had elapsed, the patient can be enrolled in this study)
4. Has taken anti-inflammatory drugs (prescribed or over-the-counter) within 14 days before the injection of the investigational product (but if the 14-day washout period had elapsed, the patient can be enrolled in this study)
5. Has taken immunosuppressive agents, including antirheumatic drugs (e.g., methotrexate or antimetabolites) within 3 months before enrollment in this study
6. With a history of drug abuse within one year prior to enrollment in this study, or showed positive results in the urine drug test or the serum alcohol test at the screening visit
7. Received an injection in the target knee within two months before enrollment in this study
8. Pregnant or breastfeeding female
9. With another joint disease apart from degenerative arthritis (e.g., systemic rheumatic inflammatory disease associated with the knee or chondrocalcinosis, hemachromatosis, inflammatory arthritis, necrosis of the trochanter, Paget's disease adjacent to a joint in the femur or tibia, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's disease in the knee joint, villonodular synovitis, synovial chondromas)
10. With an infectious disease, including HIV or hepatitis
11. With any of the following clinically significant diseases:

    * heart disease [e.g., myocardial infarction, arrhythmia, other serious heart diseases, coronary artery bypass graft (CABG)]
    * kidney disease (e.g., chronic renal failure, glomerulonephritis)
    * liver disease (e.g., liver cirrhosis, fatty liver, acute or chronic liver disease)
    * endocrine disease (e.g., hyperthyroidism, hypothyroidism, thyroiditis, diabetes insipidus, Cushing's disease)
    * insulin-dependent diabetes mellitus
    * medical history of past or current malignant tumor
    * In particular, the tumors that TissueGene-C may aggravate can be screened using the following tests:

      * Leukemia (White Blood Cell level in the hematology)
      * Osteochondroma, Chondromas, Chondroblastoma, Chondromyxoid fibroma, Chondrosarcoma (Alkaline phosphatase level in the hematology)
12. Participated in another clinical trial (using the investigational drug or a medical device) within 30 days before enrollment in this study
13. Considered inappropriate by the investigator for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-07; Primary Completion 2012-10 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Changes in IKDC Subjective Score. | Week 0 and 24
  Symptoms, sports activities, and function of the knee will be measured by the International Knee Documentation Committee (IKDC)

SECONDARY OUTCOMES:
Changes in WOMAC scores. | Week 0 and 24
  Pain, stiffness, and physical function of the knee will be measured by the Western Ontario and McMaster Universities (WOMAC)
Changes in KOOS scores. | Week 0 and 24
  Symptoms, pain and functionality of the knee joint will be evaluated via the Knee Injury and Osteoarthritis Outcome Score (KOOS)
Changes in 100 mm-VAS. | Week 0 and 24
  Pain of the knee will be measured by the 100mm Visual Analogue Scale (VAS)
MRI scan | Week 0 and 24
  Comparison of pre-procedure MRI scans to those obtained at pre-dosing and at months 6 and 12 following dosing by an independent radiographic reviewer.
Proportion of Patients Use of Rescue Medication | Week 4, 12 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Chul Won Ha, MD, PhD, Principal Investigator — Samsung Medical Center; Seong Il Bin, MD, PhD, Principal Investigator — Asan Medical Center; Myung Chul Lee, MD, PhD, Principal Investigator — Seoul National Univ. Hospital
Locations (3):
- South Korea (3):
  - Samsung Medical Center, Gangnam-gu, Seoul
  - Seoul National Univ. Hospital, Seoul
  - Asan Medical Center, Seoul